CLINICAL TRIAL: NCT06067022
Title: Temporomandibular Dysfunction in Patients With Diabetic Foot Ulcers: What Could Be the Predictors?
Brief Title: Temporomandibular Dysfunction in Patients With Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatih Enzin, assistant professor, Harran University
Other Study IDs: fatihenzin
Record Dates: First submitted 2023-09-19; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Foot Ulcer; Temporomandibular Disorder; Swallowing Disorder
Keywords: Diabetes Mellitus; Diabetic Foot Ulcer; TMJ; Oral Health; Quality of Life
MeSH Terms: conditions — Diabetic Foot; Temporomandibular Joint Disorders; Deglutition Disorders; Diabetes Mellitus | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: 42 patients with diabetic foot ulcers were included. For patients in this group, regarding diabetic foot; Sensory assessment, ulcer area and depth measurement, and diabetes management information were measured.
  Apart from these evaluations, quality of life, pain, mandibular function and oropharyngeal swallowing problems were evaluated.
  Interventions: Other: observation
- Control Group: 42 patients without diabetes were included. Patients in this group were evaluated for general health and quality of life, pain, mandibular function and oropharyngeal swallowing problems.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — Planned measurements and scales will be applied

SUMMARY:
The aim of this observational study is to investigate the effects of the type, area and duration of ulceration on jaw pain, mandibular function limitation, TMD and swallowing in individuals with diabetic foot ulcers.The main questions it aims to answer are:

* Does the change in foot structure due to diabetic foot ulcer have an effect on the temporomandibular jointand swalloving?
* What are the determinants of tempomandibular dysfunction in individuals with diabetic foot ulcers?

Participants (both groups) will be evaluated for quality of life, jaw functionality, mandibular dysfunction, oropharyngeal swallowing disorder, pain and diabetes complications.

DETAILED DESCRIPTION:
The study was planned in an observational case-control study design. 84 participants were included. Individuals who signed the Informed Consent Form were included in the study. Individuals aged between 46-80 (min-max) who were diagnosed with type 2 DM and DFU in Harran University Research and Application Hospital Endocrinology Polyclinic were included in the study group, and healthy individuals aged 37-85 (min-max) without a diagnosis of DM were included in the control group. Among the exclusion criteria for all individuals from the study, the Mini-Mental Test score should be below 24, history of psychiatric illness, cancer, neurological problems, congenital anomalies, musculoskeletal problems, having a systemic disease, facial paralysis, undergoing surgery due to spine, abdomen and/or TMJ problem and receiving any treatment related to the spine and TMJ in less than 6 months.

In the clinical evaluation of individuals with DFU about diabetes and ulcers; diabetes duration, HbA1C value, glycemic control adequacy, and peripheral arterial disease were recorded, monofilament test was performed for sensory evaluation. Ulcer type and duration were recorded, and ulcer area was measured. Individuals' quality of life was evaluated with the Ferran Powers Quality of Life Index. In the evaluation of oral health in all participants; burning mouth syndrome, dry mouth sensation, tooth loss, tooth decay, and intraoral lesions were questioned.

Participants' pain reports were evaluated using the Numerical Rating Scale (NRS).

Participants' swallowing disorders were evaluated using the Eating Assessment Tool (EAT-10).

Participants' TMJ disorders were evaluated using the Fonseca Anamnestic Index.

Participants' mandibular dysfunctions were evaluated using the Mandibular Function Disorder Questionnaire .

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Having been diagnosed with Type 2 diabetes for at least 10 years
* Not having a serious musculoskeletal, cardiac, neurological, etc. systemic disorder that may interfere with the research.
* Not having any communication problems

Exclusion Criteria:

* Having a diabetic foot ulcer
* Having a diagnosed psychiatric disease,
* Having had a temporomandibular joint operation,
* Having experienced direct or indirect trauma to the head-neck and spine area,
* Having had previous spine surgery,
* Having any mental problems,
* Having a neuromuscular problem that proves a systemic specific pathological condition such as malignant condition of the spine and/or TMJ, fracture, rheumatoid disease,
* Having had facial paralysis less than 1 year ago,
* Being diagnosed with TMD,
* Having received TMJ-related physical therapy treatment in less than 6 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Temporomandibular Dysfunction | baseline
  An umbrella term covering pain and dysfunction of the muscles of mastication (the muscles that move the jaw) and the temporomandibular joints (the joints which connect the mandible to the skull). Temporomandibular Dysfunction was assessed using the Mandibular Function Disorder Questionnaire. This valid and reliable scale evaluating mandibular dysfunction consists of two dimensions and 17 questions. The first 11 items form the Functional Capacity dimension, and the next six items form the Nutrition dimension. Each question is scored from '0' (no difficulty) to '4' (very difficult or impossible without assistance). A high total score obtained from the questionnaire indicates a high level of impairment in jaw function.

SECONDARY OUTCOMES:
Quality of life assessment | baseline
  Quality of life is an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. The participants' quality of life was evaluated using the Ferrans&Powers Quality of Life Index Diabetes Version.The Quality of Life Assessment Index consists of two parts and a total of 68 items. In the first part, in 6-point Likert order (1=not at all satisfied, 6=very satisfied) the patient's satisfaction/pleasure in various areas of life; In the second part (1=not at all important, 6=very important) the importance levels of various life areas of the patient are questioned. It is scored in the categories of health and functional capacity, socioeconomic status, psychological belief status, family status, and total quality of life. A high score indicates a good quality of life.
Swallowing Disorders | baseline
  Swallowing disorders (Dysphagia) is the medical term for swallowing difficulties. Some people with dysphagia have problems swallowing certain foods or liquids, while others can't swallow at all. Participants' swallowing disorders were evaluated using the Eating Assessment Tool (EAT-10). The scale, which evaluates the symptoms and severity of oropharyngeal swallowing disorder and is valid and reliable, consists of 10 questions. Each question is scored between '0' (no problem) and '4' (serious problem). A total score of 3 and above on the scale between 0-40 indicates a swallowing problem.
Pain assessment | baseline
  Participants' pain reports were evaluated using the Numerical Rating Scale (NRS). It is a simple, valid, and reliable method that is frequently used in measuring the severity of pain in the clinic. The participant is asked to mark a number on a 10 cm scale, on which numbers are shown in the range of "0" (no pain) to "10" (unbearable pain) for the pain he feels in the TMJ region

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Enzin, asst prof dr, Principal Investigator — Harran University
Locations (1):
- Fatih Enzin, Sanliurfa, Haliliye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided